CLINICAL TRIAL: NCT03585985
Title: Investigation of a Link Between Heart Rate Variability and Frailty in Geriatric Patients Before and After Rehabilitation With Simultaneous Evaluation of a New Camera-based Technology for Measurement of Vital Signs
Brief Title: Investigation of a Link Between Heart Rate Variability and Frailty in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 18-059
Record Dates: First submitted 2018-05-24; First posted 2018-07-13 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Fragility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 10 patients aged above 70 years with typical geriatric multimorbidity or aged above 80 years otherwise, patient in the hospital Franziskushospital Aachen on the ward of geriatric medicine
  Interventions: Procedure: Standard patient monitor; Procedure: Photoplethysmographie-Imaging (PPGI) + Infrared thermography (IRT)
- Group 2: 10 healthy elderly people above 70 years, healthy
  Interventions: Procedure: Standard patient monitor; Procedure: Photoplethysmographie-Imaging (PPGI) + Infrared thermography (IRT)

INTERVENTIONS:
Procedure: Standard patient monitor — Measurement of reference data: heart rate, heart rate variability and respiratory rate
Procedure: Photoplethysmographie-Imaging (PPGI) + Infrared thermography (IRT) — Camera-based technology for the determination of heart rate variability (PPGI) and contactless measurement of breathing rate (IRT)

SUMMARY:
The aim of this study is the evaluation of differences in heart rate variability (both time- and frequency-domain) [a]: between frail and non-frail patients and [b] at the beginning and end of a geriatric therapy which included rehabilitation components. Moreover, the suitability of new camera-based technology with regard to measurement of vital signs (heart rate, heart rate variability, respiratory rate) will be evaluated.

DETAILED DESCRIPTION:
Frailty is an important geriatric syndrome, which indicates a reduced maximum resilience of patients and their organ system against external stressors. According to Fried's classification, frailty comprises of unintentional weight loss, exhaustion, muscle weakness, slowness while walking and low levels of activity. In geriatric patients, frailty is associated with a higher mortality and morbidity. Moreover, frailty patients are more often dependent on assistance after hospitalisation than non-frailty patients.

During geriatric therapy, geriatric patients are treated with multimodal rehabilitation comprising of activating nursing, physiotherapy, occupational therapy, psychiatric and speech therapy in order to increase mobility and patients' ability to help themselves. Success of rehabilitation measures is measured using the geriatric assessment (e.g. Barthel Index, Timed up and go test, Mini-Mental State Examination, Geriatric Depression Scale, measurement of hand power) at the beginning and end of the therapy. This geriatric therapy including the named geriatric assessment is not study-specific and is not prescribed by a study protocol, but is a routine treatment for frail patients.

Apart from these routinely used tests, recent literature indicated that heart rate variability, which can be easily measured with an ECG, could be an indicator for frailty. Beyond the medical problem whether heart rate variability can be used as a surrogate parameter for frailty, this study also has a technical aspect. In biomedical engineering, non-contact monitoring of vital signs has been an important and promising development in the last decade. Therefore, this study will also investigate if camera-based technologies such as photoplethysmography imaging (PPGI) and infrared thermography (IRT) can be used in a clinical environment for non-contact measurement of vital signs (heart rate, heart rate variability, respiratory rate) in geriatric patients. In this study, monitoring (with conventional and contactless technologies) should not trigger any observable/examining effect, but is merely a means to the end of observing the already existing HRV (and other vital parameters).

ELIGIBILITY:
Inclusion Criteria:

* Group 1: aged above 70 if they have typical geriatric multimorbidity, otherwise aged above 80, patient on the geriatric ward in the hospital "Franziskhospital Aachen"
* Group 2 (Healthy volunteers): aged above 70, healthy and in good physical condition
* Written informed consent by patient / volunteer

Exclusion Criteria:

* Inability to consent
* Pace maker

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 10 patients above 70 years with frailty form the geriatric medicine ward in the Franziskushospital Aachen and 10 healthy volunteers with age above 70 years without frailty
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Link between heart rate variability and frailty | approx. 14 days (duration of geriatric complex therapy)
  heart rate variability is measured by ECG; frailty is evaluated by geriatric assessment (questionnaires)
  both investigations are not related to the study but geriatric complex therapy

SECONDARY OUTCOMES:
Correlation and precision of camera-based heart rate measurement with reference data from standard patient monitor | approx. 14 days (duration of geriatric complex therapy)
  the following devices / methods are used to record the heart rate:
  * camera-based measurement: photoplethysmography imaging (PPGI);
  * reference data: ECG
Correlation and precision of camera-based heart rate variability with reference data from standard patient monitor | approx. 14 days (duration of geriatric complex therapy)
  the following devices are used to record the heart rate variability:
  * camera-based measurement: photoplethysmography imaging (PPGI);
  * reference data: Pulsoximeter (fingerclip)
Correlation and precision of camera-based respiratory rate with reference data from standard patient monitor | approx. 14 days (duration of geriatric complex therapy)
  the following devices / methods are used to record the respiratory rate:
  * camera-based measurement: infrared thermography (IRT);
  * reference data: ECG
Development of Frailty / geriatric assessment at the beginning and end of the geriatric early-rehabilitation complex-therapy | approx. 14 days (duration of geriatric complex therapy)
  Frailty is evaluated by geriatric assessment (questionnaires)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius Bollheimer, Univ.-Prof. Dr. med., Principal Investigator — Department of Geriatrics, University Hospital RWTH Aachen Aachen, NRW, Germany, 52074 Contacts:
Locations (1):
- Department of Geriatrics, University Hospital RWTH Aachen Aachen, Aachen, North Rhine-Westphalia, Germany